CLINICAL TRIAL: NCT06173427
Title: Monitoring of Intracranial Hemorrhage in Non-severe Head Trauma Patients Hospitalized in the UHCD. Indication of a Control Imaging ?
Brief Title: Monitoring of Intracranial Hemorrhage in Non-severe Head Trauma Patients Hospitalized in the UHCD
Acronym: Head-Trauma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7492
Record Dates: First submitted 2022-11-03; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Head Trauma
Keywords: Head Trauma; Intracranial hemorrhage; Cerebral hemorrhagic lesions; Neurological monitoring; Brain scan
MeSH Terms: conditions — Craniocerebral Trauma; Intracranial Hemorrhages

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The non-neurosurgical management of post-traumatic cerebral hemorrhagic lesions is currently poorly codified. It consists of neurological monitoring for 24 to 48 hours, and the performance of an almost systematic brain scan. Anti-aggregation and anticoagulation treatments are stopped for 14 to 28 days and should be resumed according to the risk-benefit ratio and the advice of the patient's treating physicians and cardiologists.

If the bleeding lesions do not progress, the patients are allowed to return home. If the lesions progress, the patients remain hospitalized for further monitoring, a new brain scan and neurosurgical advice.

This study seeks to show that the performance of systematic brain imaging in the absence of clinical deterioration of patients admitted to the UHCD for post-traumatic intracranial hemorrhage could be avoided, and thus to administer an unnecessary dose of irradiation to the patients, and would also have a significant financial stake.

Several recent studies have shown that there is no need to perform a follow-up brain scan in the absence of neurological deterioration, even in anticoagulated patients or those on antiplatelet drugs. Despite the growing number of articles, no recommendation or consensus has been proposed.

ELIGIBILITY:
Inclusion criteria:

* Adult patient (≥18 years old)
* Admitted to Emergency department of the Strasbourg University Hospital during the year 2017 (from 01/01/2017 to 31/12/2017)
* Patient having given his consent to the reuse of his data for the purpose of this research
* Hospitalized at the University Hospital for monitoring of a post-traumatic intracranial hemorrhage

Exclusion criteria:

* Patient having expressed opposition to participate in the study
* Non-isolated cranial trauma (MVA, fall greater than 6 meters ..)
* Subject under court protection
* Subject under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient (≥18 years old) admitted to Emergency department of the Strasbourg University Hospital during the year 2017 (from 01/01/2017 to 31/12/2017)
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Retrospective description of clinical evolution of post-traumatic intracerebral hemorrhages | Through study completion, an average of 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'accueil des urgences - CHU de Strasbourg - France, Strasbourg, France